CLINICAL TRIAL: NCT01989208
Title: A Dose Escalation Study to Assess the Safety and Ability of SG1002 to Overcome Circulating Deficits in Hydrogen Sulfide Found in Heart Failure Patients
Brief Title: Assessing the Safety and Ability of SG1002 to Overcome Deficits in Hydrogen Sulfide in Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sulfagenix Australia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SG1002-001
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure
Keywords: Heart Failure; Congestive Heart Failure; Oxidative Stress; Hydrogen Sulfide
MeSH Terms: conditions — Heart Failure | interventions — sodium sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar capsule (Placebo Comparator): One normal healthy subject and two heart failure subjects will be randomized and given placebo throughout the trial period.
  Interventions: Other: Placebo
- SG1002 (Experimental): 200 mg capsule of SG1002 (alpha sulfur/sodium sulfate)
  Interventions: Other: SG1002

INTERVENTIONS:
Other: SG1002 — 200 mg capsules will be administered BID for 7 days, then doubled to 2 capsules BID for 7 days and doubled again to 4 capsules BID for the final 7 days.
  Other Names: alpha sulfur/sodium sulfate
  Arms: SG1002
Other: Placebo — 200 mg capsules containing placebo will be administered BID for 7 days, then doubled to 2 capsules BID for 7 days and doubled again to 4 capsules BID for the final 7 days.
  Arms: Sugar capsule

SUMMARY:
Patients with heart failure are reported to have lower levels of hydrogen sulfide in their blood, even though sulfur is available naturally in the diet. Hydrogen sulfide is a molecule that has been shown to have a number of beneficial effects and thus the low levels may contribute to the disease. This trial is testing whether a medical food product of synthetic sulfur molecules, SG1002, can overcome this deficit in blood levels of hydrogen sulfide.

DETAILED DESCRIPTION:
Subjects with heart failure have been shown to have a deficit in circulating hydrogen sulfide levels, which, since sulfur is not readily bioavailable and is declining in food substances, cannot be treated adequately by diet alone. This deficit in circulating hydrogen sulfide is thought to lead to increases in oxidative stress and with this, associated problems that can contribute to heart failure. This is a study to evaluate the safety and ability of multiple doses of oral SG1002 in subjects with heart failure to reverse the deficits in circulating hydrogen sulfide. The primary objective is to assess the safety and the ability of multiple doses of twice daily administration of SG1002 compared with placebo to increase circulating levels of hydrogen sulfide. Initially, a dose escalation study will be carried out for 21 days in 4 normal subjects, randomized 3:1 active:placebo. Subjects will receive a 200 mg dose BID for 7 days and in no adverse events, escalate to 400 mg for 7 days then 800 mg for 7 days. Safety parameters will be assessed for each dose, along with pharmacokinetic analysis and markers of oxidative stress and heart failure. Following completion of the normal healthy subjects, 10 heart failure subjects will be randomized 4:1 active:placebo and tested as described above.

ELIGIBILITY:
Inclusion Criteria (healthy volunteers):

* Healthy male volunteers aged between 18 and 45 years (inclusive);
* Body mass index between 19 and 30 kg/m^2 (inclusive);
* No clinically significant findings in the medical history and physical examination;
* No clinically significant laboratory values and urinalysis, unless the investigator considers any abnormality to be clinically irrelevant;
* Normal ECG, blood pressure and heart rate, unless the Investigator considers any abnormality to be not clinically significant (NCS);
* Willing to use contraception (single barrier methods); and
* Willing and able to provide written informed consent.

Exclusion Criteria (healthy volunteers):

* Have received blood products within 1 month prior to Screening;
* Have received any investigational research agent within 30 days or 5 half-lives (whichever is longer) prior to the first dose of trial medical food;
* Have received an investigational vaccine within 6 months, a live attenuated vaccine within 60 days or a registered vaccine within 30 days prior to the first dose of the trial medical food;
* Have a history of thyroidectomy or thyroid disease that required medication within the past 12 months;
* Have had serious angioedema episodes within the previous 3 years or requiring medication in the previous two years;
* Have a bleeding disorder diagnosed by a doctor (for example factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties during blood draws;
* Have a psychiatric condition that precludes compliance with the protocol, past or present psychoses, past or present bipolar disorder, or a disorder requiring lithium, within five years prior to enrolment;
* Has a history of suicide plan;
* Any clinically significant abnormality at Screening determined by medical history, physical examination, blood chemistry, haematology, urinalysis and a 12-lead ECG, or positive urine screen for drugs of abuse;
* Any other condition which in the view of the Investigator is likely to interfere with the study or put the subject at risk;
* HIV, or hepatitis B or C positive;
* Have a history of or current clinically significant gastrointestinal, hepatic, renal, cardiovascular, respiratory, endocrine, oncological, immunodeficiency, neurological, metabolic, haematological or autoimmune disorder;
* Have a history of or current tuberculosis, epilepsy, diabetes or glaucoma;
* Have clinical signs of active infection or a temperature more than 38.0°C at the time of screening. Study entry may be deferred at the discretion of the Principal Investigator;
* Have evidence of drug or alcohol abuse;
* Be unable to provide repeated blood samples without undue trauma or distress;
* Anticipate surgery within the trial period; or
* Inability to speak English (due to need to administer standardized English-language questionnaire).

Inclusion Criteria (heart failure subjects):

* Aged between 35 and 85 years (inclusive);
* Has symptomatic heart failure, with New York Heart Association (NYHA)classification of II or III;
* Ambulatory;
* Left ventricular ejection fraction less than 40%;
* Congestive heart failure has been stable for the previous 3 months (defined by no change in baseline therapy or symptoms of heart failure for the previous 3 months); and
* Willing and able to provide written informed consent.

Exclusion Criteria (heart failure subjects):

* Subject is pregnant or breastfeeding;
* If female, the subject is either post-menopausal or surgically sterilised or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide, or abstinence) from signing of the informed consent form though to the Final Visit/Early Termination Visit;
* Myocardial infarction, unstable angina, stroke, cerebrovascular accident, percutaneous coronary intervention, open heart surgery or transient ischemic attack (TIA) within 3 months prior to Screening;
* Current symptomatic hypotension (defined as systolic blood pressure (SBP) ≤ 90 mmHg or diastolic blood pressure (DBP) ≤ 40 mmHg);
* Poorly controlled hypertension (defined as SBP ≥ 160 mmHg or DBP ≥ 100 mmHg) despite therapy
* Subjects with NYHA grade IV heart failure;
* Subjects awaiting percutaneous coronary intervention or open heart surgery;
* Subjects with serious liver disease;
* Subjects with liver function test results three times the upper limit of normal.
* Any change in cardiovascular drug therapy within three months prior to randomization
* History of chronic obstructive pulmonary disease (diagnosed using GOLD criteria) or evidence of restrictive lung disease (defined as forced expiratory volume (FEV1) to forced vital capacity (FCV) ratio of > 80%);
* Poorly controlled diabetes (defined as HbA1c > 10.0 %);
* Has undergone Cardiac Resynchronisation Therapy (CRT) in the last 6 months and no planned CRT;
* Implantable cardioverter defibrillator (ICD) implant planned during the study;
* Hypersensitivity to sulfur or related compounds;
* Renal insufficiency defined as estimated Glomerular Filtration Rate (eGFR) < 30 mL/minute/1.73 m2 (Modification of Diet in Renal Disease Study MDRD) [2];
* Life expectancy less than 6 months;
* Active malignancy requiring active anti-neoplastic therapy that will, in the opinion of the investigator, interfere with study treatment or participation. (Stable basal cell skin cancer and cancers being treated solely with hormonal therapy are allowed.)
* Inability to speak English (due to need to administer standardized English-language questionnaire); or
* Any other chronic illness that may, in the opinion of the Investigator, increase the risks associated with this trial.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Lickliter, MD, PhD, Principal Investigator — Nucleus Network; Henry Krum, MBBS, PhD, Principal Investigator — The Alfred
Locations (2):
- Australia (2):
  - Alfred Health, Melbourne, Victoria
  - Nucleus Network, Melbourne, Victoria

REFERENCES:
- [Derived] Polhemus DJ, Li Z, Pattillo CB, Gojon G Sr, Gojon G Jr, Giordano T, Krum H. A novel hydrogen sulfide prodrug, SG1002, promotes hydrogen sulfide and nitric oxide bioavailability in heart failure patients. Cardiovasc Ther. 2015 Aug;33(4):216-26. doi: 10.1111/1755-5922.12128. PMID 25930144

RESULTS

PARTICIPANT FLOW:
Groups:
- Sugar Capsule: Two normal healthy subject and two heart failure subjects will be randomized and given placebo throughout the trial period.
- SG1002: 200 mg capsule of SG1002 (alpha sulfur/sodium sulfate)
  SG1002: 200 mg capsules will be administered BID for 7 days, then doubled to 2 capsules BID for 7 days and doubled again to 4 capsules BID for the final 7 days to six normal healthy subjects and six heart failure subjects.
Period: 200 mg (7 Days)
Arm/Group | Sugar Capsule | SG1002
Started | 4 | 12
Completed | 4 | 11
Not Completed | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: 400 mg (7 Days)
Arm/Group | Sugar Capsule | SG1002
Started | 4 | 11
Completed | 4 | 11
Not Completed | 0 | 0
Period: 800 mg (7 Days)
Arm/Group | Sugar Capsule | SG1002
Started | 4 | 11
Completed | 4 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SG1002: 200 mg capsule of SG1002 (alpha sulfur/sodium sulfate)
  SG1002: 200 mg capsules will be administered BID for 7 days, then doubled to 2 capsules BID for 7 days and doubled again to 4 capsules BID for the final 7 days.
  Six normal healthy subject and six heart failure subjects will be randomized and given SG1002 throughout the trial period.
- Total: Total of all reporting groups
Arm/Group | Sugar Capsule | SG1002 | Total
Number analyzed (Participants) | 4 | 12 | 16
Age, Customized [Mean (Full Range); unit: years]
  Normal Healthy Subjects | 27.0 [27 to 27] | 27.7 [25 to 34] | 27.5 [25 to 34]
  Heart Failure Subjects | 73.0 [68 to 78] | 75.5 [71 to 85] | 74.9 [68 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 4 | 10 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 11 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Australia | 4 | 12 | 16
Condition [Number; unit: participants] — Heart Failure subjects were classified as NYHA Class II (Mild symptoms, including mild shortness of breath and/or angina) and slight limitation during ordinary activity) or III (Moderate symptoms, including marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances.Comfortable only at rest.)
  participants
    Normal Healthy Subjects | 2 | 6 | 8
    Heart Failure Subjects | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: The number of subjects reporting Treatment Emergent Adverse Events at any time during the study period.
Time Frame: Following 7 days of treatment at each of three doses
Measure: Number; unit: participants
Arm/Group | Sugar Capsule | SG1002
Number analyzed (Participants) | 4 | 12
participants
  Subjects with Treatment Adverse Events | 2 | 3
  Subjects with no Treatment Emergent Adverse Events | 2 | 9

2. Secondary Outcome: Assessing Changes in Peak Hydrogen Sulfide Levels in Heart Failure Subjects Following SG1002 Administration.
Description: At the start of each dose, blood samples will be obtained and circulating hydrogen sulfide levels will be assessed over a 24 hour period to determine whether SG1002 can overcome the deficits reported in heart failure patients. Peak hydrogen sulfide levels were measured during the first 4 hours post-administration when maximum concentrations of hydrogen sulfide were reached.
Time Frame: 24 hours
Population: Heart failure subject (n=6) had baseline levels of hydrogen sulfide recorded at 0, 0.5, 1, 2, 4, 6, 12 and 24 hours after the administration of the first dose of each of the escalating doses of SG1002.
Measure: Mean (Standard Error); unit: uM
Groups:
- Baseline: Baseline levels of free hydrogen sulfide (H2S) were recorded in heart failure subjects.
- 200 mg SG1002: 200 mg capsules of SG1002 were administered BID for 7 days to heart failure subjects.
- 400 mg SG002: 400 mg capsules of SG1002 were administered BID for 7 days to heart failure subjects.
- 800 mg SG1002: 800 mg capsules of SG1002 were administered BID for 7 days to heart failure subjects.
Arm/Group | Baseline | 200 mg SG1002 | 400 mg SG002 | 800 mg SG1002
Number analyzed (Participants) | 6 | 6 | 6 | 6
uM | 0.37 (0.05) | 0.44 (0.04) | 0.50 (0.08) | 0.51 (0.09)

3. Other Pre Specified Outcome: Assessing Potential Clinical Benefits of SG1002 Administration by Analyzing BNP Levels.
Description: BNP levels were measured for the each subject prior to treatment and after 7 days on each treatment dose, thus representing a change in BNP over the 21 day treatment period. Increased BNP levels are associated with worsening heart failure.
Time Frame: 7 days at each dose.
Population: Levels of BNP were recorded at baseline and every 7 days in the placebo group or the SG1002 dose escalation group.
Measure: Mean (Standard Error); unit: pg/ml
Groups:
- Sugar Capsule: Day 0: Baseline BNP levels of the subjects receiving sugar capsules.
- Sugar Capsules: Day 7: Baseline BNP levels of the subjects receiving sugar capsules for 7 days.
- Sugar Capsules: Day 14: Baseline BNP levels of the subjects receiving sugar capsules for 14 days.
- Sugar Capsules: Day 21: Baseline BNP levels of the subjects receiving sugar capsules for 21 days.
- SG1002: Day 0: Baseline BNP levels of the subjects who were randomized to the SG1002 treatment group, prior to any drug administration.
- SG1002: Day 7: Baseline BNP levels of the subjects who were randomized to the SG1002 treatment group, following administration of 200 mg SG1002 BID for 7 days.
- SG1002: Day 14: Baseline BNP levels of the subjects who were randomized to the SG1002 treatment group, following administration of 200 mg SG1002 BID for 7 days, then 400 mg SG1002 BID for an additional 7 days.
- SG1002: Day 21: Baseline BNP levels of the subjects who were randomized to the SG1002 treatment group, following administration of 200 mg SG1002 BID for 7 days, then 400 mg SG1002 BID for an additional 7 days and then 800 mg SG1002 BID for an additional 7 days..
Arm/Group | Sugar Capsule: Day 0 | Sugar Capsules: Day 7 | Sugar Capsules: Day 14 | Sugar Capsules: Day 21 | SG1002: Day 0 | SG1002: Day 7 | SG1002: Day 14 | SG1002: Day 21
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 6 | 6 | 6 | 6
pg/ml | 85.0 (49.0) | 123.0 (72.0) | 156.5 (97.5) | 149.5 (53.5) | 77.5 (30.5) | 69.8 (26.9) | 79.0 (31.6) | 72.0 (38.7)

ADVERSE EVENTS:
Groups:
- SG1002: 200 mg capsule of SG1002 (alpha sulfur/sodium sulfate)
  SG1002: 200 mg capsules will be administered BID for 7 days, then doubled to 2 capsules BID for 7 days and doubled again to 4 capsules BID for the final 7 days.
  Six normal healthy subject and six heart failure subjects will be randomized and given placebo throughout the trial period.
Arm/Group | Sugar Capsule | SG1002
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/12
Other Adverse Events (participants affected / at risk) | 2/4 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Capsule (N=4) | SG1002 (N=12)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper Respiratory Track Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Lethargy/syncope/diahrrea (Nervous system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Technical problems in measuring free H2S levels due to sample stability made assessment of PK difficult.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No